CLINICAL TRIAL: NCT03644979
Title: Skydiving as a Model of Psychological Stress and Its Effect on Intestinal Barrier Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2017/313
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Psychological Stress Due to Skydiving

STUDY DESIGN:
Intervention Model Description: 1) Skydiving visit, 2) Negative control visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skydiving (Experimental): Tandem skydiving
  Interventions: Other: Skydiving
- Negative control (No Intervention): No skydiving

INTERVENTIONS:
Other: Skydiving — Tandem skydiving (with an experienced instructor)
  Arms: Skydiving

SUMMARY:
In this study, it will be investigated how psychological stress evoked by skydiving affects the intestinal permeability in 20 healthy subjects. Participants attend two visits: 1) Skydiving visit, 2) Negative control visit. At all visits, saliva samples, blood samples, and faecal samples are collected, and the multi-sugar permeability test is performed. In this test, participants drink a sugar solution and then collect urine for 5 and 24 h. The ratio of the sugars detected in the urine is a reflection of the intestinal permeability. Saliva samples are collected for assessment of cortisol, a stress marker. Blood and faecal samples are collected for assessment of markers of intestinal barrier function and inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to any study related procedures
2. Age > 18 till <50
3. Novice skydivers (first or second tandem jump)
4. Signed up for tandem skydive
5. Willing to abstain from probiotic products or medications known to alter gastrointestinal function throughout the study

Exclusion Criteria:

1. Abdominal surgery which might influence gastrointestinal function, except appendectomy and cholecystectomy.
2. Current diagnosis of hypertension.
3. Current diagnosis of psychiatric disease.
4. Over 100kg or with a body mass index over 35.
5. Systemic use of steroids in the last 6 weeks.
6. Use of antibiotics or antimicrobial medication in the last month.
7. Daily usage of non-steroidal anti-inflammatory drugs in the last 2 months or incidental use in the last 2 weeks prior to screening.
8. Usage of medications that could affect the barrier function, except oral contraceptives, during the 14 days prior to screening.
9. Diagnosed inflammatory gastrointestinal disease.
10. Regular use of probiotics in the last 6 weeks.
11. Smoking and/or chewable tobacco.
12. Planned changes to current diet or exercise regime.
13. Use of laxatives, anti-diarrhetics, anti-cholinergics within last 4 weeks prior to screening.
14. Use of immunosuppressant drugs within last 4 weeks prior to screening.
15. Women: Pregnancy, lactation.
16. Abuse of alcohol or drugs.
17. Any disease/condition which in the investigator's opinion could interfere with the intestinal barrier function.
18. Any clinically significant disease/condition which in the investigator's opinion could interfere with the results of the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Change in small intestinal permeability after skydiving measured as the urinary lactulose/rhamnose secretion ratio compared to negative control | 2-4 weeks

SECONDARY OUTCOMES:
Change in whole gut permeability after skydiving measured as the urinary sucralose/erythritol secretion ratio compared to negative control | 2-4 weeks
Change in colonic permeability after skydiving measured as the urinary sucralose/erythritol secretion ratio compared to negative control | 2-4 weeks
Change in gastroduodenal permeability after skydiving measured as urinary sucrose excretion | 2-4 weeks
Change in quantity of intestinal permeability markers in blood after skydiving compared to the negative control | 2-4 weeks
  fatty acid binding proteins, zonulin, claudin-3, 16S rRNA
Change in salivary cortisol levels after skydiving compared to the negative control | 2-4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

REFERENCES:
- [Derived] Roca Rubio MF, Eriksson U, Brummer RJ, Konig J. Short intense psychological stress induced by skydiving does not impair intestinal barrier function. PLoS One. 2021 Jul 8;16(7):e0254280. doi: 10.1371/journal.pone.0254280. eCollection 2021. PMID 34237102